CLINICAL TRIAL: NCT06917235
Title: Wrist and Carpal Arthrodeses. A 1-year Follow-up Study.
Status: Recruiting | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24/06567-5
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Arthrodesis; Arthrosis; Wrist Osteoarthritis
Keywords: Wrist arthrodesis; carpal arthrodesis; follow-up; surgery; fusion
MeSH Terms: conditions — Ankylosis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Arthrodesis: All patients that fit the inclusion criteria and accept the arthrodesis surgery will be followed up over the course of 1 year. The wrist and carpal arthrodesis procedures will include radioscapholunate, scaphoid-trapezium-trapezoid (STT), and four-corner arthrodeses.
  Interventions: Procedure: Wrist and carpal arthrodesis

INTERVENTIONS:
Procedure: Wrist and carpal arthrodesis — All patients that fit the inclusion criteria and accept the arthrodesis surgery will be followed up over the course of 1 year. The wrist and carpal arthrodesis procedures will include radioscapholunate, scaphoid-trapezium-trapezoid (STT), and four-corner arthrodeses.

SUMMARY:
This study at the Orthopedic Department, Drammen Hospital, examines the effectiveness and safety of various arthrodesis procedures in the wrist and carpus to relieve chronic pain and restore functional stability. Arthrodesis, which fuses two or more bones to eliminate joint mobility, is considered as a last resort when conservative treatments do not produce the desired results. The study includes patients with advanced degenerative changes, rheumatoid arthritis, or extensive injuries. Patients assessed preoperatively and postoperatively through measurements of range of motion, grip strength, and pain using various tools such as PRWHE, QuickDASH, EQ-5D-5L and NRS. The checks include X-rays and CT to evaluate healing. The data is analyzed to identify trends and factors that influence positively outcome. The follow-up takes place after 8 weeks, 3 months and 1 year postoperatively, with a focus on pain relief and functional improvement. The data are compared before and after surgery to assess the effectiveness of the intervention efficiency. The study has been applied for approval by REK, but rejected because it was assessed as a quality control project, and applied for the Data Protection Commissioner (PVO).

The data is anonymised and stored on secure servers, with switch keys stored separately. The patients give informed consent and are insured through Norwegian Patient Injury Compensation. The study seeks to improve patient care by increasing understanding of the long-term effects of osteoarthritis, including complications and secondary osteoarthritis. The results will contribute to better clinical decisions and treatments.

DETAILED DESCRIPTION:
Background Wrist and carpal arthrodesis is a well-established surgical intervention in orthopedic surgery, primarily aimed at alleviating chronic pain and restoring functional stability. The procedure involves the fusion of two or more wrist bones, eliminating joint mobility to reduce pain and improve hand function. It is generally considered a last-resort treatment when conservative measures such as medication, physical therapy, and orthotic support fail.

Candidates for arthrodesis typically include patients with severe degenerative changes, rheumatoid arthritis, post-traumatic arthritis, or significant wrist trauma, where pain and instability severely impair daily activities. The procedure aims to improve quality of life by enabling essential functions without the limitations imposed by unstable or arthritic joints.

Surgical success is measured primarily by pain relief and functional improvement. Outcomes depend on careful patient selection, precise surgical technique, and structured postoperative follow-up. Long-term studies and systematic evaluations are essential to refine treatment protocols and identify predictive factors for successful outcomes while mitigating complications such as infection, nonunion, and adjacent joint degeneration.

Objective This study evaluates the effectiveness and safety of various wrist and carpal arthrodesis procedures, including radioscapholunate, scaphoid-trapezium-trapezoid (STT), and four-corner arthrodesis, through systematic postoperative follow-up and patient outcome assessment.

Methods Inclusion Criteria:

* All patients undergoing wrist or carpal arthrodesis, regardless of the specific technique.
* Indications include advanced degenerative changes unresponsive to conservative treatment.

Preoperative Evaluation:

* Bilateral range-of-motion (ROM) assessment (flexion, extension, ulnar and radial deviation, supination, pronation).
* Imaging: X-ray (AP, lateral, oblique) and CT with 3D reconstruction.
* Grip strength measurement with a dynamometer.
* Pain assessment using the Numeric Rating Scale (NRS).
* Patient-reported outcome measures (PROMs): PRWHE, QuickDASH, and EQ-5D-5L.

Postoperative Follow-up:

* CT at 8 weeks to assess bone healing, with possible extension of cast duration and reassessment at 12 weeks.
* Referral to occupational therapy for rehabilitation.
* Follow-up at 3 months and 1 year, repeating preoperative assessments and X-ray evaluation for secondary osteoarthritis.

Data Collection & Analysis:

* Pre- vs. postoperative comparisons of pain, function, and grip strength.
* Statistical analyses: t-tests, chi-square, ANOVA, Cox regression, linear and logistic regression.
* Documentation of prior wrist surgeries and indications for arthrodesis.

Sample Size & Statistical Power: With an estimated annual inclusion of 1-5 patients and a total of 10-20 participants, statistical power is limited. The study acknowledges the risk of Type II errors due to small sample size.

Regulatory Approvals & Ethics:

* The project was reviewed by the Regional Ethics Committee (REK) and deemed a quality control study, not requiring REK approval.
* Approval from the Data Protection Officer (PVO) in Vestre Viken is pending.
* Patients will provide informed consent, ensuring voluntary participation and data confidentiality.

Data Security & Management:

* Anonymized data stored on a secure research server.
* Key-coded data stored separately in Medinsight.
* The study follows institutional guidelines for data protection and patient rights.

Expected Impact:

* Enhancing the understanding of wrist arthrodesis outcomes to improve clinical decision-making and patient care.
* Identifying factors that optimize surgical success and rehabilitation.

Timeline:

* Regulatory approvals: Winter/Spring 2024.
* Patient recruitment: Fall 2024.
* Inclusion period: 5 years.
* Follow-up completion: 1 year postoperatively for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing wrist or carpal arthrodesis, regardless of the specific technique.
* Advanced degenerative changes unresponsive to conservative treatment.

Exclusion Criteria:

* Patients who do not accept participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include all patients undergoing wrist and midcarpal arthrodesis at the Orthopedic Department, regardless of the specific type of procedure. Typical candidates are individuals with advanced degenerative changes in the radiocarpal joints who have not responded to conservative treatment modalities, such as medications, physiotherapy, or orthotic support. Indications for arthrodesis include conditions such as severe osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, or significant wrist instability following trauma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-08-15 (Estimated); Study Completion 2029-08-15 (Estimated)

PRIMARY OUTCOMES:
PRWHE (Patient-Rated Wrist/Hand Evaluation) | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  The PRWHE (Patient-Rated Wrist/Hand Evaluation) form was developed to identify the degree of pain and functional impairment of the hand and wrist. It consists of two parts, one that contains five questions that focus on pain, and one with ten questions that deal with function. The questions are answered on a numerical scale from 0 to 10, where 0 means no pain or impairment and 10 the worst pain imaginable, or inability on the part of the patient to perform a certain activity. Pain and function are weighted equally by dividing the function scores by 2, and a total sum ranging between 0 and 100 is obtained. A change of > 20 points indicates a clinically significant difference, while a change of < 10 - 12 points has little or no significance

SECONDARY OUTCOMES:
EQ-5D-5L | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  EQ-5D-5L is a standardized measurement tool to assess general health status and quality of life.
  It consists of five dimensions: mobility, independence, daily activities, pain/discomfort and anxiety/depression. Respondents assess their condition within each dimension. EQ-5D is used globally in health research, economic evaluations and public health planning.
  The EQ VAS records the respondent's overall current health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The EQ VAS provides a quantitative measure of the patient's perception of their overall health.
Patient pain | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  The NRS, or Numerical Rating Scale, is a widely used method for assessing patients' experience of pain or satisfaction.
  It consists of a scale from 0 to 10, where 0 represents "no pain" or "completely dissatisfied" and 10 indicates "worst imaginable pain" or "completely satisfied". Patients are asked to rate their pain or satisfaction level by selecting a number that best describes their current condition. The NRS is easy to administer and understand, and can be used in a number of medical and research contexts to quantify pain intensity or degree of satisfaction. This method is particularly useful for following changes in the patient's condition over time, as well as evaluating the effect of treatments or interventions. In assessments of pain and satisfaction, the person answers a standard question from the project staff. The NRS has been found to be both reliable and valid and is widely used when assessing pain and satisfaction.
Patient satisfaction | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  The NRS, or Numerical Rating Scale, is a widely used method for assessing patients' experience of pain or satisfaction. It consists of a scale from 0 to 10, where 0 represents "no pain" or "completely dissatisfied" and 10 indicates "worst imaginable pain" or "completely satisfied". Patients are asked to rate their pain or satisfaction level by selecting a number that best describes their current condition. The NRS is easy to administer and understand, and can be used in a number of medical and research contexts to quantify pain intensity or degree of satisfaction. This method is particularly useful for following changes in the patient's condition over time, as well as evaluating the effect of treatments or interventions. In assessments of pain and satisfaction, the person answers a standard question from the project staff. The NRS has been found to be both reliable and valid and is widely used when assessing pain and satisfaction.
QuickDASH | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  QuickDASH (the shortened version of the Disabilities of the Arm, Shoulder, and Hand questionnaire) is a tool developed to assess the level of function and symptoms in arms, shoulders and hands in people with various conditions.
  It is a shortened version of the original DASH questionnaire and consists of 11 questions that focus on the physical function and symptom burden related to upper extremity musculoskeletal disorders. QuickDASH is designed to be simple and quick to administer, making it a practical tool for clinicians and researchers to measure patient health status and monitor changes over time. It can be used in a variety of settings, including clinical practice, research and population studies, and it supports treatment planning and outcome measurement for individuals with arm, shoulder and hand problems.
  The total score is scaled between 0 (no disability) and 100 (maximum symptoms and disability), with an average value of 10 among the general population of the United States.
Grip strength | Baseline, then at follow-ups at 3 and 12 months following the surgery, a total of 1 year.
  Grip strength is measured by means of a dynamometer. The dynamometer apparatus measures grip strength in kilograms of resistance by squeezing an adjustable (for hand size) stirrup. The higher the number of kilograms measured, the stronger the the grip strength.

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Drammen Sykehus, Drammen
  - Vestre Viken HF, Drammen

IPD SHARING:
Plan to Share IPD: No
Not allowed by Regional Ethics Committee according to